CLINICAL TRIAL: NCT06099262
Title: GenPMTO - Adaptation and Feasibility Study
Brief Title: GenPMTO Evaluation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Behavioural Insights Team (Other)
Collaborators: Implementation Sciences International, Inc (Unknown); Barnardos (Unknown)
Responsible Party: Principal Investigator, Tom McBride, Director, The Behavioural Insights Team
Other Study IDs: 2023056
Record Dates: First submitted 2023-09-26; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Violence; Emotional Adjustment; Parenting; Parent-Child Relations
Keywords: young people; youth violence; parenting programme

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Tower Hamlets 1: Delivering the GenPMTO programme to one group of caregivers within the Tower Hamlets borough.
  Interventions: Behavioral: GenPMTO
- Tower Hamlets 2: Delivering the GenPMTO programme to a second group of caregivers within the Tower Hamlets borough.
  Interventions: Behavioral: GenPMTO
- Brent 1: Delivering the GenPMTO programme to one group of caregivers within the Brent borough.
  Interventions: Behavioral: GenPMTO
- Brent 2: Delivering the GenPMTO programme to a second group of caregivers within the Brent borough.
  Interventions: Behavioral: GenPMTO
- Barking & Dagenham 1: Delivering the GenPMTO programme to one group of caregivers within the Barking & Dagenham borough.
  Interventions: Behavioral: GenPMTO
- Barking & Dagenham 2: Delivering the GenPMTO programme to a second group of caregivers within the Barking & Dagenham borough.
  Interventions: Behavioral: GenPMTO

INTERVENTIONS:
Behavioral: GenPMTO — GenPMTO is a parenting programme which involves trained practitioners using active teaching approaches (such as group problem-solving, role-play, and video modelling) to support caregivers in using positive parenting strategies at home. The programme is designed to improve parenting practices, as well as a range of outcomes for young people, including improving academic performance, reducing school exclusions, and reducing offending and criminal behaviour. The version of the programme investigated in this project is delivered to groups of parents.

SUMMARY:
This project is a multi-stage evaluation of GenPMTO (Generation Parent Management Training - Oregon Model). GenPMTO is a parenting programme which involves trained practitioners using active teaching approaches (such as group problem-solving, role-play, and video modelling) to support caregivers in using positive parenting strategies at home. The programme is designed to improve parenting practices, as well as a range of outcomes for young people, including improving academic performance, reducing school exclusions, and reducing offending and criminal behaviour. The version of the programme investigated in this project is delivered to groups of parents.

DETAILED DESCRIPTION:
This project represents the first attempt to deliver and evaluate GenPMTO in the UK. To do so, the Ending Youth Violence Lab, at the Behavioural Insights Team, is conducting a multi-stage evaluation, involving delivering the intervention across three London boroughs, with a focus on caregivers of 8-14-year-old children and young people (CYPs), who are identified to have risk factors associated with involvement in violence.

To design this project, the Lab has collaborated with two partners. The first is ISII (Implementation Sciences International, Inc.), a research-based, non-profit organisation based in the USA, which implements the GenPMTO programme, in partnership with the programme developers. ISII also trains community practitioners in its use across the world. The second partner is Barnardo's, the UK's largest children's charity, and the delivery partner for the project.

This entry refers to the first 2 stages of the project, which will run concurrently:

Stage 1 - Adaptation and training

* The purpose of this Stage is to prepare for initial delivery and the feasibility testing of delivery, by making any adaptations that may be necessary for the UK context and beginning practitioner training.
* The research objectives of this Stage firstly focus on identifying whether the programme may require adaptations to fit into the UK context and identifying and justifying appropriate adaptations. Secondly, the investigators want to identify whether sufficient numbers of practitioners can be recruited and trained within the budget of the project, and to identify the optimal approach to recruitment and training of future practitioner cohorts to allow delivery at a larger scale.

Stage 2 - Feasibility study

The purpose of this Stage is to understand the feasibility of delivering GenPMTO to the caregivers of children who have been identified as being at risk of violence, through testing recruitment, retention, fidelity, etc. The investigators will also conduct further adaptation to the programme as necessary, responding to what we learn from practitioners and caregivers who have experienced the programme for the first time.

The specific research objectives here focus on:

* Feasibility - Can Barnardo's recruit and retain caregivers of children who meet inclusion criteria and are at risk of youth violence, and deliver the programme withfidelity?
* Acceptability - Is the GenPMTO programme seen as acceptable and valuable by caregivers and practitioners in a UK context?
* Evaluability - Firstly, is there sufficient demand and capacity to deliver GenPMTO at a scale required for a randomised control trial? Secondly, is it feasible to collect outcome data from participants, which would support robust outcome data collection procedures during a pilot and/or efficacy trial?

This will involve delivering the programme in 3 London boroughs, and collecting a range of survey data and conducting qualitative interviews with caregivers and with practitioners to explore the above questions. The investigators will collect pre- and post-programme outcome data using a range of self-report measures, to explore the potential for future robust evaluation (rather than to assess programme impact).

ELIGIBILITY:
Inclusion Criteria - Caregivers are eligible to participate in the feasibility study (including receiving GenPMTO) if they:

* Have a child or young person (CYP) between the ages of 8-14.
* Are the primary caregiver (i.e. spend the most time with the CYP and are available to care for them).
* Live within one of the boroughs in which GenPMTO is being delivered (during the feasibility study).

And, if one of or more of the following is present:

* CYPs have engaged in criminal behaviour, such as breaking the law or "offending behaviour" - for both non-violent and violent crimes.
* CYPs have engaged in violent and challenging behaviour (including within the home, e.g. against parents and/or siblings).
* CYPs have been reported as bullying other individual(s) in or outside of school settings.
* CYPs have low attendance at school (<50% within the last academic year).
* CYPs have been excluded from school within the last academic year.
* CYPs are engaged in substance abuse/misuse (e.g. drugs, alcohol)
* CYPs are at risk of involvement by gangs.
* CYPs are at risk of exploitation, or negative influence, by criminal peers.
* CYPs have a sibling(s) that has entered into the criminal justice system.

Exclusion Criteria - Caregivers will be excluded from the feasibility study it at least any of the following are present:

* Caregiver(s) have received a parenting programme in the last two months, or are currently receiving one.
* Caregiver(s) and CYP does not have working proficiency in English, such that participation in GenPMTO and research activities would be unfeasible.
* Family has plans to move out of the borough within the 10-14 week delivery timeline, and thus may not be available for full delivery of GenPMTO during the feasibility study phase.
* Severe developmental delay for caregiver or CYP which may prevent caregiver from attending GenPMTO delivery sessions, implementing GenPMTO parenting strategies, or participating in evaluation.
* Caregiver(s) and/or CYPs are actively homicidal, suicidal or psychotic.
* Problem sexual behaviour is the central behavioural concern for child/young person.
* Significant child protection concern (i.e. basic needs of children are not being met by caregivers.

Ages: 8 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Caregivers of young people aged 8-14, who have been identified as being at risk of committing violent acts and/or entering into the criminal justice system.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of practitioners recruited to deliver GenPMTO | Prior to delivery of the intervention
  This will involve calculating, as a percentage, the number of recruited practitioners, compared to the target.
Proportion of practitioners enrolled in training to deliver GenPMTO | Throughout delivery of the intervention - approximately 5 months
  This will involve calculating, as a percentage, the number of practitioners enrolled in training, compared to the target.
Number of referrals received for caregivers to receive GenPMTO | Prior to delivery of the intervention
  This will involve identifying the total count of referrals received during the feasibility study, as well the mean and standard deviation of monthly referral totals across the feasibility study.
Proportion of referred caregivers deemed eligible for GenPMTO | Prior to delivery of the intervention
  This will involve calculating, as a percentage, the number of caregivers deemed eligible for GenPMTO, compared to to the total number of referred caregivers.
Proportion of eligible caregivers who are offered GenPMTO who accept this offer (take-up of services) | Prior to delivery of the intervention
  This will involve calculating, as a percentage, the number of caregivers who consent to take part in the feasibility study, compared to to the total number of caregivers who are considered eligible to receive and are offered the programme.
Retention / drop-out rates of caregivers receiving GenPMTO | Throughout delivery of the intervention - approximately 5 months
  This will involve calculating, as a percentage, the number of caregivers who complete a program, compared to the total number of caregivers who consent to receiving GenPMTO
Retention / drop-out rates of practitioners delivering GenPMTO | Throughout delivery of the intervention - approximately 5 months
  This will involve calculating, as a percentage, the number of practitioners who have completed relevant training and are able to deliver GenPMTO, compared to the total number of practitioners who were enrolled in training.
Attendance rate at GenPMTO sessions | Throughout delivery of the intervention - approximately 5 months
  This will involve calculating, as a percentage, the number of caregivers who attended each GenPMTO session, compared to the number of caregivers who were expected (i.e. based on caregiver take-up/enrollment) to attend these sessions, as well the mean and standard deviation across the feasibility study.
Caregivers' perception of the quality of the content and delivery | Within 1 month after the end of the intervention
  This will involve calculating the mean and standard deviation of scores, based on a short feedback survey.
Programme dosage data | Throughout delivery of the intervention - approximately 5 months
  This will involve calculating the mean percentage of actual content delivered in GenPMTO sessions to a cohort of caregivers, compared to the amount of planned content to be delivered.
Ratings of practitioner fidelity | Throughout delivery of the intervention - approximately 5 months
  This will involve calculating the mean of practitioners' fidelity scores whilst delivering a full GenPMTO programme. Fidelity is measured using the Fidelity of Implementation (FIMP) Rating System system (expert assessment of videotaped sessions). Each session is assessed on a 9 point scale (1 referring to 'needs work', and 9 referring to 'good work').
Parenting approach | Within 1 month after the end of the intervention
  Parenting Practices Interview (self-reported measure)
  This is a 64 item measure, with responses measured on a 1-7 Likert scale. Total scores range from 64 to 448, with higher scores indicating improved parenting practices.
Parental self-efficacy | Within 1 month after the end of the intervention
  Parental Locus of Control-Short Form Revised (self-report)
  This is a 24 item measure, with responses measured on a 1-5 Likert scale. Total scores range from 24 to 120, with higher scores indicating greater parental self-efficacy.
Behavioural problems | Within 1 month after the end of the intervention
  Strengths and Difficulties Questionnaire (parent report of child)
  The overall (five-subscale) SDQ score ranges from 0 to 50, with a higher score indicating abnormal behaviours. The Total Difficulties score ranges from 0 to 40. The externalising score ranges from 0 to 20 and is the sum of the conduct and hyperactivity scales. The internalising score ranges from 0 to 20 and is the sum of the emotional and peer problems scales. Higher scores indicate abnormal behaviours.
Behavioural problems | Within 1 month after the end of the intervention
  Eyberg Child Behaviour Inventory (parent report of child)
  7-point Likert scale, from 1 ('Never Occurs') to 7 ('Always Occurs') and a Yes/No Problem scale. Individual Intensity Score items are summed up, with resultant scores ranging from 36 to 252. For each item, the parents' response regarding whether the behaviour is a problem for them ('Yes' = 1 , 'No' = 0) is also summed to create the Problem Score, ranging from 0 to 36.
Offending behaviour - Variety | Within 1 month after the end of the intervention
  Young people are asked to report on offending behaviours they have participated in.
  Variety of delinquency score:
  Sum the number of items the respondent answers 'yes' to:
  Yes = 1 No = 0
  Produces a score that ranges from 0-19, where a higher score indicates a higher variety of delinquency.
Offending behaviour - Volume | Within 1 month after the end of the intervention
  Self-reported delinquency scale (child self-report measure)
  Young people are asked to report on offending behaviours they have participated in.
  Volume of delinquency score:
  Summing the point values when respondents report a number of times. Point values are assigned as follows:
  Once = 1 Twice = 2 3 times = 3 4 times = 4 5 times = 5 Between 6 and 10 times = 6 More than 10 times = 11
  Produces a score that ranges from 0 to 11 for each delinquent behaviour, where a higher score indicates a higher volume of delinquency
Victimisation | Within 1 month after the end of the intervention
  Victimisation sub-scale of the Problem Behaviour Frequency Scale (child self-report measure)
  Produces a score ranging from 6-36 achieved by summing scores of the two subscales, where a higher score indicates a higher frequency of problem behaviours

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - London Borough of Barking and Dagenham, London
  - London Borough of Brent, London
  - London Borough of Tower Hamlets, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project description and study protocol — https://www.bi.team/projects/genpmto/

DOCUMENTS (1):
  • Study Protocol (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT06099262/Prot_000.pdf